CLINICAL TRIAL: NCT01408745
Title: Multicenter Controlled Study on the Safety and Efficacy of Sternal Closure With STERNUMFIX in Patients With High Risk
Brief Title: Sternal Closure With STERNUMFIX in Patients With High Risk
Acronym: STEPHIX
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: terminatedd due to insufficient recruitment
Sponsor: Aesculap AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AAG-G-H-0802
Record Dates: First submitted 2011-07-19; First posted 2011-08-03 (Estimated); Last update posted 2015-04-14 (Estimated); Status verified 2015-04

CONDITIONS: Sternum Wound Infection; Nonunion of Fracture of Sternum
Keywords: medical device; sternal closure; sternotomy; dehiscence; sternal wound healing; randomized trial; steel wire

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sternumfix (Experimental): sternotomy closure with Sternumfix
  Interventions: Device: Sternumfix
- Steel wire (Active Comparator): sternotomy closure with steel wire
  Interventions: Procedure: steel wire

INTERVENTIONS:
Device: Sternumfix — sternotomy closure with Sternumfix
  Arms: Sternumfix
Procedure: steel wire — sternotomy closure with steel wire
  Arms: Steel wire

SUMMARY:
The primary objective is to establish if the SternumFix System improves sternal closure. The study should test the hypothesis that in a high risk patient population with increased risk for the development of sternal wound complications SternumFix will reduce the incidence of sternal healing complications. The control group will be treated with wire cerclage, the standard method of sternal closure.

ELIGIBILITY:
Inclusion:

* Patients undergoing elective cardiac surgery with a median sternotomy
* Age >18 years
* Male and female sex
* Informed consent
* Patients with high risk for sternal wound complications

Patients are designated as high risk patients if they have either:

* one or more major risk factors or
* four or more minor risk factors.

Major risk factors are:

* Obesity: BMI > 30.
* Diabetes: intake of oral anti-diabetic drugs and/or insulin at time of surgery.
* COPD: history of chronic coughing plus expectoration for at least 3 months by at least two consecutive years, plus evidence of restrictive pattern at spirometry.
* Planned BITA: bilateral use of thoracic artery
* Age > 75 years

Minor risk factors are:

* History of smoking;(minimum of 1 year of history of smoking)
* Hyperlipoproteinaemia (as stated in the patient data)
* Planned surgery is a CABG
* Patient is on dialysis
* Repeat sternotomy
* Left ventricular ejection fraction < 30% (as stated in the patient data)
* Male sex

Exclusion:

* Active infection
* Participation in a pharmaceutical clinical study or any trial with interfering endpoints within the last 30 days
* Pregnancy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 166 (Actual)
Dates: Start 2008-06; Primary Completion 2012-08 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
cumulative three-months incidence of re-operation rates due to sternal instability or infection for patients with SternumFix in comparison to sternal fixation with wires in a high risk patient population | within three months

SECONDARY OUTCOMES:
Adverse event rate. Postoperative chest pain. Length of postoperative hospital stay. Blood loss within the first 12 hours p.o. Duration of the sternal fixation. | within 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Roland Hetzer, Prof., Principal Investigator — Direktor der Klinik für Herz-, Thorax- und Gefäßchirurgie des DHZB
Locations (4):
- Germany (3):
  - Kerckhoff Klinik, Bad Nauheim
  - Deutsches Herzzentrum Berlin, Berlin
  - Evangelisch-Freikirchliches Krankenhaus und Herzzentrum Brandenburg in Bernau, Bernau
- University Hospital Zürich, Zurich, Switzerland